CLINICAL TRIAL: NCT06232161
Title: Retrospective,2-Year Post-Trial Follow-up Study of Sustained and Rebound Effect of Red-light Therapy for Myopia in Ningbo.
Brief Title: Sustained Effect of Red-light Therapy for Myopia Control: A 2-Year Post-Trial Follow-up Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Airdoc Technology Co., Ltd. (Industry)
Collaborators: Ningbo Eye Hospital (Other)
Responsible Party: Principal Investigator, Qiu Kaikai, Myopia control officer, Ningbo Eye Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ningbo EYE Hospital
Record Dates: First submitted 2024-01-20; First posted 2024-01-30 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Myopia
Keywords: myopia, red-light therapy
MeSH Terms: conditions — Myopia | interventions — Therapeutics; Lasers; Low-Level Light Therapy; Eyeglasses

STUDY DESIGN:
Intervention Model Description: The first 12-month follow-up were parallel of two groups: treatment group and control group with randomized and single blind; While the second 12-month follow-up were chosen to be in the treatment group or in the control group depended on the willingness of red-light therapy from both patients and their family.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- red-light therapy group (Experimental): The red-light therapy group would be treated with red-light therapy twice daily including the single focus spectacles during the follow-up.
  Interventions: Device: Red-light therapy device; Device: Spectacles
- control group (Other): The control group including both the stopping red-light therapy group from the first 12 months (who obtained red-light therapy but stopped during the second 12-month follow-up) and those never use red-light therapy.
  Interventions: Device: Spectacles

INTERVENTIONS:
Device: Red-light therapy device — Red-light therapy was performed with a low-intensity laser (LD-A, Jilin LD Optoelectronics Technology, Jilin, China) with an irradiance of 0.35 ± 0.02 mW/cm2, a wavelength of 650 nm ± 10 nm, and illumination of approximately 400 lux on average.
  Other Names: Repeated low-level red-light (RLRL) therapy; Low intensity red light (laser) therapy; Photobiomodulation therapy (PBM) therapy
  Arms: red-light therapy group
Device: Spectacles — Single focus spectacles, that is to say, wearing glasseses with minus power lens

SUMMARY:
To evaluate the long-term efficacy and safety of red-light therapy for myopia control over 2 years, and the potential rebound effect after treatment cessation.

The Chinese myopic children who originally completed the one-year randomised controlled trial in the previous study were enrolled. Children continued or started to daily usage of red-light therapy were defined as the RL group, while those who stopped using red-light therapy and switched to single-vision spectacles (SVS) as well as those who continued to keep single-vision spectacles in the second year were both regarded as the SVS group. Red-light therapy was provided by an at-home desktop light device emitting red-light of 650 nm and was administered for 3 min at a time, twice a day. Changes in axial length (AL) and cycloplegic spherical equivalence refraction (SER) are to be measured and compared as well as the adverse effects including the rebound effect.

Red-light therapy has emerged as a novel myopia control treatment modality recently. A 12-month randomised controlled trial (RCT) conducted by our research team was thought to be earlier to evaluate the treatment of myopic children using red-light therapy. The trial demonstrated that PBM therapy was effective on myopia control, reducing axial elongation and spherical equivalence refraction (SER) progression 103% and 127% compared with single vision spectacle (SVS) over a 12-month period, respectively. The promising efficacy of red-light therapy has been further confirmed in other studies. In addition, satisfactory user acceptability and no unrecovered functional and structural damages were observed.

Myopia generally progresses throughout childhood and hence a study duration of 1 year is not sufficient to widely adopt the red-light therapy as a treatment strategy for myopia control. The sustainability of treatment efficacy, rebound phenomenon upon cessation of treatment, and potential risks and adverse effects in myopic children with longer-term PBM therapy, remain to be fully elucidated.

Thus, the aims of this post-trial follow-up study were to invite the participants to come back for a 24-month visit and to investigate the long-term efficacy and safety of continued red-light therapy as well as the potential rebound effect following red-light treatment cessation.

DETAILED DESCRIPTION:
Interventions and visits All spectacle lenses were made for single focus with full correction for each subject as the first intervention throughout the whole procedure for both groups. PBM therapy was performed with a low-intensity laser (LD-A, Jilin LD Optoelectronics Technology, Jilin, China) with an irradiance of 0.35 ± 0.02 mW/cm2, a wavelength of 650 nm ± 10 nm, and illumination of approximately 400 lux on average at the first 12 month. At the second 12 months, non-randomized cohorts continued according to the willing to use the device from both groups. Once decided, those usage would be followed up for another 12 months for tracking the change of axial length as well as the change of refractive error. All the adverse effects and any harms are encouraged to report during the next 12 months' study.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of myopia;
2. Ages of 9~13 years old;
3. Must be with best corrected visual acuity ≥20/25 (decimal record);
4. Must be the subject in the previous study of 12-month red-light therapy of myopia;

Exclusion Criteria:

1. Clinical diagnosis of glaucoma or retinal lesions;
2. Clinical diagnosis of optic media lesions (e.g., central thick corneal scars, cataract);
3. Clinical diagnosis of optic nerve dysfunction;
4. Clinical diagnosis of amblyopia;
5. Must be eligible for follow-up.

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2020-05-13 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of axial length (mm) with the measurement of device named by IntraOcular Lens Master(IOLmaster 500) | 12-month
  The change of axial length (mm) from the 24 months and 12 months from the baseline for each subject; The right eye were considered for the comparison between groups.
  The change value is recorded of the average from 5 values at the same follow-up

SECONDARY OUTCOMES:
Change of refractive error (D) with cycloplegic refraction with the same autorefractor | 12-month
  The change of refractive error (D) from the follow-up of each 12-month from the baseline. The right eye were considered for the comparison

CONTACTS AND LOCATIONS:
Overall Officials: LEI ZHOU, M.D., Study Chair — Ningbo Eye Hospital
Locations (1):
- Ningbo Eye Hospital, Ningbo, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Zhou L, Tong L, Li Y, Williams BT, Qiu K. Photobiomodulation therapy retarded axial length growth in children with myopia: evidence from a 12-month randomized controlled trial evidence. Sci Rep. 2023 Feb 27;13(1):3321. doi: 10.1038/s41598-023-30500-7. PMID 36849626
- See also: The first 12-month follow-up report of PBM therapy — https://pubmed.ncbi.nlm.nih.gov/36849626/